CLINICAL TRIAL: NCT00005421
Title: Blood Pressure Tracking--Childhood to Young Adulthood
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4339; R03HL048289 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To extend analyses of blood pressure (BP) tracking to a period that spanned childhood and young adulthood. Data were used from the same cohort of 339 children who had been followed for nine to twelve years in a previous study.

DETAILED DESCRIPTION:
BACKGROUND:

Blood pressure measurements in childhood and young adulthood are less predictive of future levels than those taken in middle age. In part, this may be due to the fact that within-person variability appears to make up a larger proportion of total variability in childhood than adulthood. Previous work on an NHLBI supported grant indicated that repeated blood pressure measurements and visits led to higher childhood tracking correlations over a period of three years.

DESIGN NARRATIVE:

Follow-up data were used as well as multiple visits which reduced the large within-person variability of blood pressure measurements and improved the tracking correlations. In addition, 'true' or 'corrected' tracking correlations were provided by eliminating the effects of random measurement error. The effects were examined of time-varying covariates on both the observed and true tracking correlations. Besides computing tracking correlations, predictive values were computed for young adult blood pressure given childhood levels. This was the probability that a young adult's true blood pressure was above a specific cutpoint conditional on childhood blood pressure. These values were validated using data from the Fels Longitudinal Study, which included serial blood pressure measurements over the age range in the study. The prediction models were also derived including terms for covariates such as age, sex, height and weight. From these models nomograms were constructed which were useful to physicians for prognostic purposes. Thus, because of the unique multiple-visit approach used in these data, the effect of random measurement error was eliminated. These methodologic improvements strengthened the usefulness of blood pressure screening in childhood to detect those at high risk of developing hypertension.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1995-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Cook — Brigham and Women's Hospital

REFERENCES:
- [Background] Cook NR, Gillman MW, Rosner BA, Taylor JO, Hennekens CH. Prediction of young adult blood pressure from childhood blood pressure, height, and weight. J Clin Epidemiol. 1997 May;50(5):571-9. doi: 10.1016/s0895-4356(97)00046-2. PMID 9180649
- [Background] Cook NR. Estimating predictive values for blood pressure measurements from multivariate regression models with covariates. Stat Med. 1996 Oct 15;15(19):2013-28. doi: 10.1002/(SICI)1097-0258(19961015)15:193.0.CO;2-Y. PMID 8896136
- [Background] Gillman MW, Cook NR. Blood pressure measurement in childhood epidemiological studies. Circulation. 1995 Aug 15;92(4):1049-57. doi: 10.1161/01.cir.92.4.1049. PMID 7641339
- [Background] Cook NR, Cohen J, Hebert PR, Taylor JO, Hennekens CH. Implications of small reductions in diastolic blood pressure for primary prevention. Arch Intern Med. 1995 Apr 10;155(7):701-9. PMID 7695458
- [Background] Gillman MW, Cook NR, Rosner B, Evans DA, Keough ME, Taylor JO, Hennekens CH. Identifying children at high risk for the development of essential hypertension. J Pediatr. 1993 Jun;122(6):837-46. doi: 10.1016/s0022-3476(09)90005-1. PMID 8501557